CLINICAL TRIAL: NCT06776900
Title: Video-assisted Fiberoptic Intubation in Lateral Versus Supine Position in Pediatrics Undergoing Non-head-and-neck Surgery: a Randomized Controlled Non-inferiority Trial
Brief Title: Fiberoptic Intubation in Lateral Versus Supine Position in Pediatrics Undergoing Non-head-and-neck Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS-526-2024
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Video-assisted; Head and Neck Surgery; Intubation
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine group (Active Comparator): the patient will be kept in supine position with the head placed neutrally and a roll under the shoulders
  Interventions: Procedure: Supine position
- Lateral group (Active Comparator): the patient will be positioned in the lateral position with head and neck physiologically aligned with head positioner. The dependent leg will be flexed at the hip and knee and the upper leg will be straight with a pillow between both legs
  Interventions: Procedure: Lateral position

INTERVENTIONS:
Procedure: Supine position — An assistant will be asked to hold the tongue in protrusion using a gauze held by a Magill forceps (preventing it from falling backwards). The operator will introduce the bronchoscope orally allowing its advancement till it reaches the laryngeal inlet. The glottic view will be graded from 1 (larynx is only seen) to 5 (the epiglottis down folded and larynx cannot be seen directly) (10).
  The scope will be manipulated to pass between the 2 vocal cords, and then advanced till the carina is seen to glide the suitable ETT into the trachea. Once the ETT is connected to the mechanical ventilator, chest auscultation and capnography waves will be used to confirm a successful intubation.
  At any intubation attempt where SpO2 reaches 90%, the procedure will be suspended and mechanical ventilation via a facemask applied till SpO2 of 100% achieved.
  Arms: Supine group
Procedure: Lateral position — An assistant will be asked to hold the tongue in protrusion using a gauze held by a Magill forceps (preventing it from falling backwards). The operator will introduce the bronchoscope orally allowing its advancement till it reaches the laryngeal inlet. The glottic view will be graded from 1 (larynx is only seen) to 5 (the epiglottis down folded and larynx cannot be seen directly) (10).
  The scope will be manipulated to pass between the 2 vocal cords, and then advanced till the carina is seen to glide the suitable ETT into the trachea. Once the ETT is connected to the mechanical ventilator, chest auscultation and capnography waves will be used to confirm a successful intubation.
  At any intubation attempt where SpO2 reaches 90%, the procedure will be suspended and mechanical ventilation via a facemask applied till SpO2 of 100% achieved.
  Arms: Lateral group

SUMMARY:
Fiberoptic intubation was first described in the late 1960s and has since become an effective and well-established technique for airway management in awake, sedated, and anesthetized patients. This technique is especially useful in patients with known or suspected difficult airways such as those with limited mouth opening, reduced neck mobility, cervical spine injury, obesity, or an elevated risk for aspiration. The benefits of fiberoptic intubation also include fewer complications such as tooth injury and oropharyngeal bleeding; and the opportunity for optimal positioning of double-lumen tubes in patients undergoing thoracic surgery.

Anesthesiologists may be confronted with situations in which patients in a lateral position during surgery experience an accidental loss of airway patency. Intubation with direct laryngoscopy is more challenging and time-consuming in patients in the lateral position than in the supine position, particularly when there is an abrupt loss of airway patency, as demonstrated by prior research. These observations suggest that there is an unmet need for a reliable method of airway management for patients in the lateral position. Although the airway is of a larger caliber and ventilation renders less peak and better oxygenation when patients are in the lateral position, glottic view was unfavorable for intubation when Macintosh direct laryngoscope was used in this position. This could be the reason why such a procedure is unfamiliar in anesthesia even when it is the most needed in special situations. Flexible fiberoptic intubation in lateral position would be convenient in emergency situations like accidental extubation during surgery or inadequate regional anesthesia requiring general anesthesia. Flexible fiberoptic intubation in lateral position would be of significant assistance in neurosurgical patients especially those with occipital lesions and patients with difficult airway scores with limited mouth opening or neck extension.

After thorough literature review, we found that studies comparing flexible video-assisted fiberoptic intubation in the lateral versus supine position in pediatrics are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-10 years old.
* Both genders.
* ASA physical status I and II.
* Elective non-head-and-neck surgeries.

Exclusion Criteria:

* Refusal of patients.
* Head and neck surgeries or with history of previous ones.
* Head, neck and lung congenital deformities or pathologies.
* Patients with expected difficult intubation (based on examination).
* Patients with neuromuscular disorders.
* Hypoxia: defined as low oxygen saturation (SpO2) ≤ 95% on room air.
* Trauma patients or patients requiring emergency procedures.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-01-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | 5 minutes from endoscope insertion between teeth
  time from inserting the endoscope between teeth in the first intubation attempt, till successful display of end tidal carbon dioxide (ETCO2) waveform on capnography

SECONDARY OUTCOMES:
Rate of successful intubation at first attempt. | 5 minutes from endoscope insertion between teeth
  each intubation trial will be labelled as successful from first, second or third attempt or failed
Overall number of intubation attempts | 5 minutes from endoscope insertion between teeth
  each intubation trial will be labelled as successful from first, second or third attempt or failed
Incidence of complications | 10 minutes from endoscope insertion between teeth
  Oesophageal intubation, Lip, tongue or dental injury, Oxygen desaturation (SpO2 ≤ 92%), or Bronchospasm
Oxygen saturation | 5 minutes from endoscope insertion between teeth
  just before and immediately after successful intubation

CONTACTS AND LOCATIONS:
Overall Officials: Mariam KE Mohammed, MBBCh, Principal Investigator — Cairo University; Karim KF Girgis, M.D., Study Chair — Cairo University; Sherif M Soaida, M.D., Study Director — Cairo University; Kareem MA Nawwar, M.D., Study Director — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt